CLINICAL TRIAL: NCT00712725
Title: A Phase IIb, Multicenter, Randomized, Double-blind, Placebo-Controlled Dose-finding Study of MK3207 in the Treatment of Acute Migraine
Brief Title: MK3207 for Treatment of Acute Migraines (3207-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3207-005; 2008_536
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — 2-(8-(3,5-difluorophenyl)-10-oxo-6,9-diazaspiro(4.5)dec-9-yl)-N-(2'-oxo-1,1',2',3-tetrahydrospiro(indene-2,3'-pyrrolo(2,3-b)pyridin)-5-yl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 1 (Experimental): MK3207- 2.5 mg
  Interventions: Drug: MK3207- 2.5 mg
- 2 (Experimental): MK3207- 5 mg
  Interventions: Drug: MK3207- 5 mg
- 3 (Experimental): MK3207- 10 mg
  Interventions: Drug: MK3207- 10 mg
- 4 (Experimental): MK3207- 20 mg
  Interventions: Drug: MK3207- 20 mg
- 5 (Experimental): MK3207- 50 mg
  Interventions: Drug: MK3207- 50 mg
- 6 (Experimental): MK3207- 100 mg
  Interventions: Drug: MK3207- 100 mg
- 7 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: MK3207- 2.5 mg — Arm 1: MK3207 2.5 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 1
Drug: MK3207- 5 mg — Arm 2: MK3207 5 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 2
Drug: MK3207- 10 mg — Arm 3: MK3207 10 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 3
Drug: MK3207- 20 mg — Arm 4: MK3207 20 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 4
Drug: MK3207- 50 mg — Arm 5: MK3207 50 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 5
Drug: MK3207- 100 mg — Arm 6: MK3207 100 mg taken after migraine onset.
  Other Names: MK3207
  Arms: 6
Drug: Comparator: placebo (unspecified) — Placebo taken after migraine onset.
  Arms: 7

SUMMARY:
The purpose of the study is to demonstrate the effectiveness and appropriate dosage level of MK3207 in the treatment of acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women from 18 to 65 years of age
* 1+ year history of migraine that typically last from 4 to 72 hours if untreated
* Had from 2 to 8 moderate or severe migraine attacks per month in the last 2 months
* Not pregnant or planning to become pregnant in next 6 months

Exclusion Criteria:

* Pregnant or breast-feeding, or planning to become pregnant in next 6 months
* Cannot distinguish migraine attacks from tension type headaches
* Migraines are mild or resolve without medication in less than 2 hours
* More than 15 headache-days per month or have taken medication on more than 10 days per month in the last 3 months
* Basilar type or hemiplegic migraine headaches
* More than 50 years old when migraines began
* History of cardiovascular disorder within last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Hewitt DJ, Aurora SK, Dodick DW, Goadsby PJ, Ge YJ, Bachman R, Taraborelli D, Fan X, Assaid C, Lines C, Ho TW. Randomized controlled trial of the CGRP receptor antagonist MK-3207 in the acute treatment of migraine. Cephalalgia. 2011 Apr;31(6):712-22. doi: 10.1177/0333102411398399. Epub 2011 Mar 7. PMID 21383045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 47 neurological and general research centers worldwide (19 in the United States and 28 internationally). The primary therapy period was between 2-Jul-08 to 16-Jan-09.
Pre-assignment Details: Participants were assessed using the protocol inclusion and exclusion criteria at Visit 1 and, if eligible, were randomized at the same visit.
Groups:
- Placebo: Placebo; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 2.5 mg: MK3207 2.5 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 5 mg: MK3207 5 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 10 mg: MK3207 10 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 20 mg: MK3207 20 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 50 mg: MK3207 50 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 100 mg: MK3207 100 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
- MK3207 200 mg: MK3207 200 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
Period: Overall Study
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Started | 169 | 39 | 57 | 84 | 86 | 84 | 83 | 74
Completed | 140 (The "Not Completed" patients discontinued prior to receiving study medication.) | 33 (The "Not Completed" patients discontinued prior to receiving study medication.) | 47 (The "Not Completed" patients discontinued prior to receiving study medication.) | 67 (The "Not Completed" patients discontinued prior to receiving study medication.) | 67 (The "Not Completed" patients discontinued prior to receiving study medication.) | 68 (The "Not Completed" patients discontinued prior to receiving study medication.) | 61 (One patient received study drug. The remaining patients discontinued prior to receiving study drug.) | 63 (The "Not Completed" patients discontinued prior to receiving study medication.)
Not Completed | 29 | 6 | 10 | 17 | 19 | 16 | 22 | 11
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 1 | 1 | 2 | 2 | 3 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 3 | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 2
Not completed — Lack of Qualifying Event | 16 | 2 | 6 | 8 | 11 | 13 | 11 | 6
Not completed — Protocol Specified Criteria | 3 | 0 | 1 | 2 | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 2.5 mg: MK3207 2.5 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 5 mg: MK3207 5 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 10 mg: MK3207 10 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 20 mg: MK3207 20 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 50 mg: MK3207 50 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 100 mg: MK3207 100 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- MK3207 200 mg: MK3207 200 mg; one orally administered dose to treat a single moderate-to-severe migraine headache.
  The participants reported in the Baseline Characteristics are randomized participants that received study treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg | Total
Number analyzed (Participants) | 140 | 33 | 47 | 67 | 67 | 68 | 62 | 63 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.2) | 43.3 (10.5) | 43.4 (11.1) | 44.1 (10.0) | 44.1 (11.3) | 42.2 (10.8) | 42.2 (10.9) | 40.5 (10.7) | 42.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 27 | 40 | 62 | 54 | 62 | 52 | 54 | 476
  Male | 15 | 6 | 7 | 5 | 13 | 6 | 10 | 9 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 4 | 4 | 4 | 10 | 13 | 9 | 10 | 69
  Not Hispanic or Latino | 125 | 29 | 43 | 63 | 57 | 55 | 53 | 53 | 478
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 132 | 32 | 46 | 62 | 63 | 64 | 59 | 59 | 517
  Black | 5 | 0 | 1 | 3 | 1 | 2 | 2 | 3 | 17
  Asian | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 6
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Multi-Racial | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Study Region [Number; unit: Participants]
  United States | 66 | 14 | 22 | 30 | 39 | 45 | 34 | 20 | 270
  Ex-United States | 74 | 19 | 25 | 37 | 28 | 23 | 28 | 43 | 277

OUTCOME MEASURES:

1. Primary Outcome: Pain Freedom (PF)
Description: Reduction of a Grade 2 or 3 severity migraine at baseline to Grade 0 at 2 hours postdose.
  Rating of Headache Severity (Scale from Grade 0 to 3):
  * Grade 0: No pain
  * Grade 1: Mild pain
  * Grade 2: Moderate pain
  * Grade 3: Severe pain
Time Frame: 2 hours postdose
Population: Full Analysis Set (FAS), which included all randomized participants who administered study treatment, had both a baseline severity measurement and at least one postdose efficacy measurement prior to or including the 2-hour time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 44 | 63 | 63 | 65 | 59 | 58
Participants | 13 | 4 | 5 | 16 | 12 | 14 | 14 | 21
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p < 0.001, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with PF at 2 hours postdose as the dependent variable; Model adjusted for geographic region (US, ex-US), baseline severity (moderate, severe), treatment and age (continuous), using identity link function

2. Secondary Outcome: Pain Relief (PR)
Description: Reduction of a Grade 2 or 3 severity migraine at baseline to mild or no pain (Grade 1 or 0) at 2 hours postdose.
  Rating of Headache Severity (Scale from Grade 0 to 3):
  * Grade 0: No pain
  * Grade 1: Mild pain
  * Grade 2: Moderate pain
  * Grade 3: Severe pain
Time Frame: 2 hours postdose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 44 | 63 | 63 | 65 | 59 | 58
Participants | 48 | 15 | 19 | 36 | 36 | 41 | 31 | 40
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p < 0.001, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with binary response PR at 2 hours postdose as the dependent variable; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Absence of Photophobia
Description: Absence of photophobia at 2 hours postdose as recorded by patient on paper diary.
Time Frame: 2 hours postdose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 44 | 63 | 63 | 65 | 59 | 58
Participants | 51 | 10 | 15 | 32 | 27 | 32 | 26 | 33
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p < 0.001, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with Absence of Photophobia at 2 hours postdose as the dependent variable; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Absence of Phonophobia
Description: Absence of phonophobia at 2 hours postdose as recorded by patient on paper diary.
Time Frame: 2 hours postdose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 44 | 63 | 63 | 65 | 59 | 58
Participants | 57 | 12 | 18 | 35 | 35 | 38 | 31 | 37
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p < 0.001, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with Absence of Phonophobia at 2 hours postdose as the dependent variable; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Absence of Nausea
Description: Absence of nausea at 2 hours postdose as recorded by patient on paper diary.
Time Frame: 2 hours postdose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 43 | 63 | 63 | 65 | 59 | 58
Participants | 79 | 19 | 25 | 44 | 42 | 44 | 41 | 45
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p = 0.007, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with Absence of Nausea at 2 hours postdose as the dependent variable; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Sustained Pain Freedom (SPF)
Description: Pain freedom (Grade 0) at 2 hours postdose, with no administration of any rescue medication and no occurrence thereafter of a mild/moderate/severe headache during the 2 to 24 hours after dosing with study medication.
Time Frame: 2-24 hours postdose
Population: Full Analysis Set (FAS), which included all randomized participants who met the FAS criteria for PF at 2 hours postdose, and who, between 2-24 hours posedose, either 1) did not have PF at any time, 2) used rescue, or 3) answered the 24 hour recurrence question.
Measure: Number; unit: Participants
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Number analyzed (Participants) | 133 | 32 | 44 | 63 | 63 | 65 | 59 | 58
Participants | 10 | 4 | 2 | 13 | 10 | 12 | 12 | 17
Statistical Analysis 1: Comparison: Placebo vs MK3207 2.5 mg vs MK3207 5 mg vs MK3207 10 mg vs MK3207 20 mg vs MK3207 50 mg vs MK3207 100 mg vs MK3207 200 mg; Test type: Superiority or Other; p < 0.001, Generalized linear regression model — p-value constructed from trend test of dose response, by testing the slope of the MK3207 dose covariate (all dose groups included) in a generalized linear regression model with binary response SPF 2-24 hours postdose as the dependent variable; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Patients were assessed for AEs from V1 (Pre-treatment Screening/Randomization) through 14 days after the dose of study medication was taken. AEs that occurred prior to administration of study medication were not included in AE summaries.
Description: Every patient is counted a single time for each applicable specific adverse event.
  Patients in population are patients who took at least one tablet of the study medication.
  Placebo is the pooled arm of all matching placebo doses.
Arm/Group | Placebo | MK3207 2.5 mg | MK3207 5 mg | MK3207 10 mg | MK3207 20 mg | MK3207 50 mg | MK3207 100 mg | MK3207 200 mg
Serious Adverse Events (participants affected / at risk) | 1/142 | 0/32 | 0/47 | 1/66 | 0/67 | 0/68 | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 20/142 | 10/32 | 18/47 | 9/66 | 14/67 | 16/68 | 17/62 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=142) | MK3207 2.5 mg (N=32) | MK3207 5 mg (N=47) | MK3207 10 mg (N=66) | MK3207 20 mg (N=67) | MK3207 50 mg (N=68) | MK3207 100 mg (N=62) | MK3207 200 mg (N=63)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0/0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=142) | MK3207 2.5 mg (N=32) | MK3207 5 mg (N=47) | MK3207 10 mg (N=66) | MK3207 20 mg (N=67) | MK3207 50 mg (N=68) | MK3207 100 mg (N=62) | MK3207 200 mg (N=63)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 3 | 1 | 2 | 4 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 2 | 3 | 5 | 3 | 5 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 2 | 2 | 2 | 4 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 4 | 2 | 2 | 2 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 2 | 0 | 2 | 3 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.